CLINICAL TRIAL: NCT05111769
Title: Preliminary Study on the Clinical Effect of Recombinant Human Brain Natriuretic Peptide on Sepsis Complicated With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEPSIS-HF
Record Dates: First submitted 2021-09-30; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Sepsis
Keywords: sepsis; Heart Failure; AKI
MeSH Terms: conditions — Sepsis; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rhBNP in the treatment of sepsis complicated with heart failure (Experimental): Recombinant human brain natriuretic peptide (rhBNP) on sepsis complicated with heart failure
  Interventions: Drug: Recombinant human brain natriuretic peptide
- Conventional treatment group (No Intervention): Do not use recombinant human brain natriuretic peptide (rhBNP) to treat sepsis with heart failure

INTERVENTIONS:
Drug: Recombinant human brain natriuretic peptide — 1. To determine the effect of rhBNP on hemodynamics in sepsis based on PiCCO hemodynamic monitoring; 2. To collect and sort out the relevant data to determine the effects of rhBNP on cardiac function and kidney function, including cardiac ultrasound, kidney blood flow index and related laboratory tests. 3. To determine the effect of rhBNP on the final prognosis of patients, including ICU mortality and hospital mortality, ICU time, hospital stay, ventilator use time, kidney replacement therapy time, vasoactive drug dosage and time.
  Arms: rhBNP in the treatment of sepsis complicated with heart failure

SUMMARY:
The investigators intend to conduct clinical studies to determine the efficacy of rhBNP in the treatment of septic related dysfunction and kidney dysfunction

DETAILED DESCRIPTION:
Sepsis is one of the common critical diseases in ICU with high mortality. Septic shock patients are often accompanied by multiple organ dysfunction (MODS), of which more than 50% of patients with varying degrees of myocardial injury.The investigators hope to find a drug with a protective effect on cardiac function and kidney function, so as to treat sepsis more effectively in the treatment of sepsis.

Recombinant human brain natriuretic peptide (rhBNP) was approved by FDA in 2001 for the treatment of acute decompensated heart failure.These effects play a role in the protection of cardiac and kidney function, and have achieved good results in patients with cardiac insufficiency and AKI caused by cardiac surgery.

The investigators are going to carry out related research from the following aspects: 1. To determine the effect of rhBNP on hemodynamics in sepsis based on PiCCO hemodynamic monitoring; 2. To collect and sort out the relevant data to determine the effects of rhBNP on cardiac function and kidney function, including cardiac ultrasound, kidney blood flow index and related laboratory tests. 3. To determine the effect of rhBNP on the final prognosis of patients, including ICU mortality and hospital mortality, ICU time, hospital stay, ventilator use time, kidney replacement therapy time, vasoactive drug dosage and time.

ELIGIBILITY:
Inclusion Criteria:

* sepsis complicated with heart failure（Diagnosed by sepsis 3.0）
* Heart failure: BNP rises by 600 pg/ml
* Age>=18 years old

Exclusion Criteria:

* Hemodynamically unstable
* Pregnant
* Disagree with comprehensive and active life support treatment
* coronary heart disease, myocardial infarction, and cardiac insufficiency
* chronic renal insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
the effects of rhBNP(recombinant human brain natriuretic peptide) on cardiac function | 72 hours after rhBNP
  The decreasing trend of NTproBNP(N-terminal pro-B-type natriuretic peptide)
PiCCO hemodynamic monitoring in recombinant human brain natriuretic peptide group | 72 hours after recombinant human brain natriuretic peptide
  The improvement degree of cardiac index in recombinant human brain natriuretic peptide group

SECONDARY OUTCOMES:
ICU mortality and hospital mortality | One month after entering ICU
  Comparison between rhBNP group and control group
Mechanical ventilation time after entering ICU | 72 hours after recombinant human brain natriuretic peptide
  Comparison between rhBNP group and control group

CONTACTS AND LOCATIONS:
Locations (1):
- Ju Minjie, Shanghai, Shanghai Municipality, China